CLINICAL TRIAL: NCT04006457
Title: A PHASE 3 OPEN-LABEL, MULTI-CENTER, LONG-TERM STUDY INVESTIGATING THE SAFETY AND EFFICACY OF PF-06651600 IN ADULT AND ADOLESCENT PARTICIPANTS WITH ALOPECIA AREATA
Brief Title: Long-Term PF-06651600 for the Treatment of Alopecia Areata
Acronym: ALLEGRO-LT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B7981032; 2023-509801-59-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Results first posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Alopecia Areata
Keywords: Alopecia; Alopecia Areata; Alopecia totalis; Alopecia universalis; Hair loss; JAK inhibitor; PF-06651600; Ritlecitinib
MeSH Terms: conditions — Alopecia Areata; Alopecia; Alopecia universalis | interventions — PF-06651600; Tetanus Toxoid; Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment sequence 1 (Experimental): Participants who did not previously receive study intervention in either study B7931005 or B7981015 will receive 200 milligrams (mg) PF-06651600, given as four 50 mg tablets once daily (QD) for 1 month, followed by 50 mg PF-06651600 tablet or capsule given QD for 59 months.
  Patients participating in the vaccine sub-study will receive the 2 vaccines or one of the 2 vaccines at the vaccine sub-study Day 1, which will occur at a scheduled study visit on or after the Month 9 visit and prior to or on the Month 56 visit of the main B7981032 study.
  Interventions: Drug: PF-06651600; Biological: Tetanus and diphtheria toxoids and acellular pertussis (Tdap) vaccine; Biological: Meningococcal (groups A, C, W-135 and Y [ACWY]) oligosaccharide diphtheria CRM197 conjugate vaccine
- Treatment sequence 2 (Experimental): Participants who previously received study intervention in either study B7931005 or B7981015 will receive 50 mg PF-06651600 tablet or capsule given QD for 59 months.
  Patients participating in the vaccine sub-study will receive the 2 vaccines or 1 of the 2 vaccines at the vaccine sub-study Day 1, which will occur at a scheduled study visit on or after the Month 6 visit and prior to or on the Month 56 visit of the main B7981032 study.
  Interventions: Drug: PF-06651600; Biological: Tetanus and diphtheria toxoids and acellular pertussis (Tdap) vaccine; Biological: Meningococcal (groups A, C, W-135 and Y [ACWY]) oligosaccharide diphtheria CRM197 conjugate vaccine

INTERVENTIONS:
Drug: PF-06651600 — 50 mg oral tablets/capsules
Biological: Tetanus and diphtheria toxoids and acellular pertussis (Tdap) vaccine — Single intramuscular injection administered to patients participating in the vaccine sub-study
Biological: Meningococcal (groups A, C, W-135 and Y [ACWY]) oligosaccharide diphtheria CRM197 conjugate vaccine — Single intramuscular injection administered to patients participating in the vaccine sub-study

SUMMARY:
This is a global Phase 3 study to evaluate the safety and effectiveness of an investigational study drug (called PF-06651600) in adults and adolescents (12 years and older) who have alopecia areata. Eligible patients from the prior studies B7931005 (NCT02974868) and B7981015 (NCT03732807) will have an opportunity to enroll as well as patients who have not previously participated in either of these studies. The study is open-label and all patients entering the study will receive active study drug.

A sub-study of approximately 60 adult patients who are participating in the B7981032 study will be conducted at select sites in the US, Australia and Canada. The sub-study will evaluate the immune response to tetanus and meningococcal vaccines in patients who have received a minimum of 6 months of 50 mg PF-06651600.

ELIGIBILITY:
Inclusion Criteria-

For de novo participants and participants from Study B7931005 and B7981015 with >30 days between first visit in B7981032 and last dose in the prior study:

* Clinical diagnosis of alopecia areata (AA) with no other cause of hair loss. Androgenetic alopecia coexistent with AA is allowed.
* De novo participants >=12 to <18 years of age: >=50% terminal hair loss of the scalp due to AA, including alopecia totalis and alopecia universalis
* De novo participants >=18 years of age and participants from Study B7931005 or B7981015 with >30 days between first visit in B7981032 and last dose in the prior study: >=25% terminal hair loss of the scalp due to AA, including alopecia totalis and alopecia universalis
* No evidence of terminal scalp hair regrowth within 6 months (de novo only)
* Current episode of terminal scalp hair loss <=10 years (de novo only)

Exclusion Criteria-

For de novo participants and participants from Study B7931005 and B7981015 with >30 days between first visit in B7981032 and last dose in the prior study:

* Hearing loss with progression over previous 5 years, or sudden hearing loss, or middle or inner ear disease, or other auditory condition that is considered acute, fluctuating or progressive
* History of or current malignancies with the exception of adequately treated or excised non metastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ
* History of a single episode of disseminated herpes zoster or disseminated herpes simplex, or a history of more than one episode of localized, dermatomal herpes zoster
* Infection requiring hospitalization, or parenteral antimicrobial therapy within 6 months prior to Day 1

Exclusion criteria for all participants:

- Participants who have previously taken Janus kinase (JAK) inhibitors other than PF-06651600 must have received the last dose >12 weeks prior to the screening visit

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1052 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2026-01-23 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (143):
- United States (47):
  - The University of Alabama at Birmingham Hosptial Outreach Lab, Birmingham, Alabama
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - The University of Alabama at Birmingham, Department of Dermatology, Birmingham, Alabama
  - Mosaic Dermatology, Beverly Hills, California
  - Univ of California, Irvine, Dermatology Clinical Research Center, Irvine, California
  - Dermatology Specialists Inc., Murrieta, California
  - University of California, San Francisco, San Francisco, California
  - Kaiser Permanente Clinical Trials Unit, San Francisco, California
  - Southern California Dermatology, Inc., Santa Ana, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Colorado Hospital Clinical and Translational Research Center, Aurora, Colorado
  - University of Colorado Hospital Outpatient Pavilion, Aurora, Colorado
  - Yale School of Medicine, Yale Center for Clinical Investigations, New Haven, Connecticut
  - Medstar Georgetown University Hospital - Department of Otolaryngology, Washington D.C., District of Columbia
  - Medstar Georgetown University Hospital-Dept of Otolaryngology, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Medstar Georgetown University Hospital - Department of Pediatrics, Washington D.C., District of Columbia
  - Siperstein Dermatology Group, Boynton Beach, Florida
  - Park Avenue Dermatology, Orange Park, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Velocity Clinical Research - Boise, Meridian, Idaho
  - Northwestern Medical Group, Chicago, Illinois
  - Northwestern Medicine Diagnostic Testing Center, Chicago, Illinois
  - Northwestern Medicine, Chicago, Illinois
  - Northwestern Memorial Hospital Investigational Drug Service Pharmacy, Chicago, Illinois
  - Summit Dermatology and Aesthetic Surgery (in c/o TrialSpark, Inc), Oakbrook Terrace, Illinois
  - NorthShore University HealthSystem Dermatology Clinical Trials Unit, Skokie, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Medstar Georgetown University Hospital - Department of Dermatology, Chevy Chase, Maryland
  - Massachusetts General Hospital - Clinical Unit for Research Trials in Skin (CURTIS), Boston, Massachusetts
  - University of Minnesota Clinical Research Unit (CRU), Minneapolis, Minnesota
  - University of Minnesota Lillehei Clinical Research Unit (LCRU), Minneapolis, Minnesota
  - University of Minnesota Medical Center, Investigational Drug Services Attn: Darlette Luke, Minneapolis, Minnesota
  - Skin Specialists, PC (Schlessinger MD), Omaha, Nebraska
  - Schweiger Dermatology, P.C., Verona, New Jersey
  - NYU School of Medicine, The Ronald O. Perelman Department of Dermatology, New York, New York
  - Pura Dermatology (in c/o TrialSpark, Inc), New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - UNC CTRC, Chapel Hill, North Carolina
  - UNC Dermatology and Skin Cancer Center, Chapel Hill, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Vital Prospects Clinical Research Institute, P.C., Tulsa, Oklahoma
  - Oregon Medical Research Center, Portland, Oregon
  - The University of Texas Health Science Center at Houston, Bellaire, Texas
  - Tamjidi Skin Institute (in c/o TrialSpark, Inc), Vienna, Virginia
- Argentina (2):
  - CINME Centro de Investigaciones Metabolicas, CABA, Buenos Aires
  - Psoriahue Medicina Interdisciplinaria, CABA
- Australia (7):
  - Premier Specialists Pty Ltd, Kogarah, New South Wales
  - St George Dermatology & Skin Cancer Centre, Kogarah, New South Wales
  - The Skin Centre, Benowa, Queensland
  - Veracity Clinical Research Pty Ltd, Woolloongabba, Queensland
  - Skin Health Institute, Carlton, Victoria
  - Sinclair Dermatology, East Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Canada (11):
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - Eastern Canada Cutaneous Research Associates Ltd., Halifax, Nova Scotia
  - Sudbury Skin Clinique, Greater Sudbury, Ontario
  - Guenther Research Inc, London, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - The Centre for Clinical Trials, Oakville, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - York Dermatology Clinic and Research Centre, Richmond Hill, Ontario
  - Research Toronto, Toronto, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
  - Centre de Recherche Dermatologique du Quebec metropolitain (CRDQ), Québec, Quebec
- Chile (4):
  - Centro Medico Skin Med, Santiago, LAS Condes
  - Centro Internacional de Estudios Clinicos - CIEC, Santiago, Recoleta
  - Clinica Dermacross S.A., Santiago, Vitacura
  - Medical Skin Center, Viña del Mar
- China (8):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The University of Hong Kong - Shenzhen Hospital, Shenzhen, Guangdong
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - Ruijin Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou, Zhejiang
- Colombia (3):
  - Fundacion Centro de Investigacion Clinica CIC, Medellín, Antioquia
  - Fundacion Hospitalaria San Vicente de Paul, Medellín, Antioquia
  - Centro de Investigacion en Reumatologia y Especialidades Medicas S.A.S, CIREEM S.A.S, Bogota D.C.
- Czechia (4):
  - DERMAMEDICA s.r.o., Náchod
  - Fakultni nemocnice Olomouc, Olomouc
  - Clintrial s.r.o., Prague
  - Sanatorium profesora Arenbergera, Prague
- Germany (6):
  - Fachklinik Bad Bentheim, Bad Bentheim
  - Emovis GmbH, Berlin
  - Universitaetsklinikum Erlangen, Erlangen
  - University Hospital Frankfurt, Frankfurt am Main
  - University Hospital Schleswig-Holstein, Lübeck
  - University Hospital Muenster, Münster
- Japan (7):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Tohoku University Hospital, Sendai, Miyagi
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Juntendo Tokyo Koto Geriatric Medical Center, Koto-ku, Tokyo
  - Kyorin University Hospital, Mitaka-shi, Tokyo
  - Osaka Metropolitan University Hospital, Osaka
  - Tokyo Medical University Hospital, Tokyo
- Mexico (2):
  - Sociedad de Metabolismo y Corazon S.C., Veracruz
  - Hospital D Maria, Veracruz
- Poland (12):
  - Twoja Przychodnia SCM, Szczecin, West Pomeranian Voivodeship
  - McBk S.C., Grodzisk Mazowiecki
  - Centermed Krakow Sp.z o.o., Krakow
  - Dermoklinika Centrum Medyczne s.c. M.Kierstan, J. Narbutt, A. Lesiak, Lodz
  - Dermedic Jacek Zdybski, Ostrowiec Świętokrzyski
  - RCMed Oddzial Warszawa, Warsaw
  - Magdalena Opadczuk Carpe Diem Centrum Medycyny Estetycznej, Warsaw
  - ETG Warszawa, Warsaw
  - Royalderm Agnieszka Nawrocka, Warsaw
  - EMC Instytut Medyczny S.A. Przychodnia przy ul. Lowieckiej we Wroclawiu, Wroclaw
  - Cityclinic Przychodnia Lekarsko Psychologiczna Matusiak Spółka Partnerska, Wroclaw
  - Centrum Medyczne OPOROW, Wroclaw
- Russia (9):
  - State Budgetary Healthcare Institution "Chelyabinsk Regional Clinical Dermatovenerologic Dispensary", Chelyabinsk
  - University Clinic of Kirov SMU, Kirov
  - FSBEI HE Russian University of Medicine of the MoH of Russia, Moscow
  - Federal State Autonomous Institution "National Medical Research Centre of Children's' Health", Moscow
  - State Budgetary Institution of the Rostov Region "Dermatovenerologic Dispensary", Rostov-on-Don
  - Limited Liability Company "Centre Vitiligo" ("Centre Vitiligo" LLC), Saint Petersburg
  - Limited Liability Company "Pierre Volkenshtein Skin Diseases Clinic", Saint Petersburg
  - Saint Petersburg State Budgetary Healthcare Institution "Dermatovenerologic Dispensary No. 10 -, Saint Petersburg
  - State Autonomous Healthcare Institution of the Yaroslavl Region "Clinical Emergency Hospital, Yaroslavl
- South Korea (2):
  - Pusan National University Hospital, Busan
  - Seoul National University Hospital, Seoul
- Spain (7):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario La Paz: Servicio de Farmacia, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario y Politecnico La Fe, Valencia
- Taiwan (6):
  - Chung-Shan Medical University Hospital, Taichung, R.o.c.
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Medical Foundation Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taipei Medical University-Shuang Ho Hospital, Ministry of Health and Welfare, New Taipei City
  - National Taiwan University Hospital, Taipei
  - Chang Gung Medical Foundation Linkou Chang Gung Memorial Hospital, Taoyuan
- United Kingdom (6):
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire
  - University Hospitals Sussex NHS Foundation Trust (UHSussex), Brighton
  - NHS Greater Glasgow and Clyde, Queen Elizabeth University Hospital, Glasgow
  - Guy's and St Thomas Hospitals NHS Foundation Trust, St Thomas Hospital, London
  - Guy's and St Thomas' Hospitals NHS Foundation Trust, St Thomas' Hospital, London
  - Guy's and St Thomas' Hospitals NHS Foundation Trust, Guy's Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Ueki R, Mizuashi M, Harada K, Zhang X, Wu W, Chung WH, Kwon O, Luo X, Basey V, Wolk R, Shi N, Fujita K, Shen Y, Hirose T. Efficacy and Safety of Ritlecitinib in the Asian Subpopulation of the ALLEGRO-2b/3 and ALLEGRO-LT Clinical Studies for Alopecia Areata. J Dermatol. 2026 Feb 6. doi: 10.1111/1346-8138.70154. Online ahead of print. PMID 41645877
- [Derived] Ishowo-Adejumo R, Zareba A, Wajsbrot D, Wolk R. Responses to Tetanus and Meningococcal Vaccines in Patients with Alopecia Areata Treated with Ritlecitinib. Dermatol Ther (Heidelb). 2026 Jan 24. doi: 10.1007/s13555-025-01648-z. Online ahead of print. PMID 41579233
- [Derived] King B, Mirmirani P, Lo Sicco K, Ramot Y, Sinclair R, Asfour L, Ezzedine K, Paul C, Ohyama M, Edwards RA, Bonfanti G, Kerkmann U, Wajsbrot D, Ishowo-Adejumo R, Zwillich SH, Lejeune A. Patterns of clinical response in patients with alopecia areata treated with ritlecitinib in the ALLEGRO clinical development programme. J Eur Acad Dermatol Venereol. 2025 Jun;39(6):1163-1173. doi: 10.1111/jdv.20547. Epub 2025 Feb 17. PMID 39962358
- [Derived] Tziotzios C, Sinclair R, Lesiak A, Mehlis S, Kinoshita-Ise M, Tsianakas A, Luo X, Law EH, Ishowo-Adejumo R, Wolk R, Sadrarhami M, Lejeune A. Long-term safety and efficacy of ritlecitinib in adults and adolescents with alopecia areata and at least 25% scalp hair loss: Results from the ALLEGRO-LT phase 3, open-label study. J Eur Acad Dermatol Venereol. 2025 Jun;39(6):1152-1162. doi: 10.1111/jdv.20526. Epub 2025 Jan 23. PMID 39846397
- [Derived] Piliang M, Soung J, King B, Shapiro J, Rudnicka L, Farrant P, Magnolo N, Piraccini BM, Luo X, Wolk R, Woodworth D, Schaefer G, Lejeune A. Efficacy and safety of the oral Janus kinase 3/tyrosine kinase expressed in hepatocellular carcinoma family kinase inhibitor ritlecitinib over 24 months: integrated analysis of the ALLEGRO phase IIb/III and long-term phase III clinical studies in alopecia areata. Br J Dermatol. 2025 Jan 24;192(2):215-227. doi: 10.1093/bjd/ljae365. PMID 39432738
- [Derived] King B, Soung J, Tziotzios C, Rudnicka L, Joly P, Gooderham M, Sinclair R, Mesinkovska NA, Paul C, Gong Y, Anway SD, Tran H, Wolk R, Zwillich SH, Lejeune A. Integrated Safety Analysis of Ritlecitinib, an Oral JAK3/TEC Family Kinase Inhibitor, for the Treatment of Alopecia Areata from the ALLEGRO Clinical Trial Program. Am J Clin Dermatol. 2024 Mar;25(2):299-314. doi: 10.1007/s40257-024-00846-3. Epub 2024 Jan 23. PMID 38263353
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7981032

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consisted of Main study and vaccine sub-study. A total of 1052 participants were enrolled in the Main study and a total of 17 participants who received at least 6 months of study treatment in the main study were enrolled in the vaccine sub-study. Results are reported at primary completion date (PCD).
Groups:
- Main Study: Ritlecitinib 200 mg/ 50 mg QD (de Novo Participants): Participants with a clinical diagnosis of alopecia areata (AA) received ritlecitinib (PF-06651600) 200 milligrams (mg) once daily (QD) for 4 weeks followed by 50 mg ritlecitinib QD for 35 months during treatment period 1. After completion of treatment period 1, participants not continuing to treatment period 2 entered a follow-up period of 4 weeks. Participants from countries where ritlecitinib was not commercially available continued to receive 50 mg ritlecitinib QD in treatment period 2 for a maximum of 24 months or until availability of commercial product in their country, or until the sponsor terminated the study in that country, whichever occurred first. Participants who permanently discontinued study treatment entered an Observation Period where they completed the scheduled study visits for approximately 2 years or until study end, whichever occurred first.Adolescent participants who did not achieve a SALT score of 20 or less by Month 6 were required to discontinue their participation in the study.
- Main Study: Ritlecitinib 50 mg QD (Roll-over Participants): Participants with a clinical diagnosis of AA who received ritlecitinib in studies B7931005 (NCT02974868) and B7981015 (NCT03732807) received 50 mg ritlecitinib QD for 36 months in treatment period 1. After completion of treatment period 1, participants not continuing to treatment period 2 entered a follow-up period of 4 weeks. Participants from countries where ritlecitinib was not commercially available continued to receive 50 mg ritlecitinib QD in treatment period 2 for a maximum of 24 months or until availability of commercial product in their country, or until the sponsor terminated the study in that country, whichever occurred first. Participants who permanently discontinued study treatment entered an Observation Period where they completed the scheduled study visits for approximately 2 years or until study end, whichever occurred first. Adolescent participants who did not achieve a SALT score of 20 or less by Month 6 were required to discontinue their participation in the study.
- Vaccine Sub-study: Tdap With or Without Meningococcal ACWY Vaccine: Participants who received at least 6 months of treatment with ritlecitinib 50 mg QD in the Main study continued to receive the study treatment in the main study while participating in vaccine sub-study. Participants were administered a single dose of Tetanus and Diphtheria Toxoids and Acellular Pertussis (Tdap) vaccine with or without a single dose of meningococcal ACWY vaccine intramuscularly on Day 1 of the sub-study.
Period: Main Study: Treatment Period 1
Arm/Group | Main Study: Ritlecitinib 200 mg/ 50 mg QD (de Novo Participants) | Main Study: Ritlecitinib 50 mg QD (Roll-over Participants) | Vaccine Sub-study: Tdap With or Without Meningococcal ACWY Vaccine
Started | 449 | 603 | 0
Treated | 447 | 603 | 0
Completed | 289 | 332 | 0
Not Completed | 160 | 271 | 0
Not completed — Adverse Event | 26 | 36 | 0
Not completed — Death | 1 | 1 | 0
Not completed — Lack of Efficacy | 27 | 79 | 0
Not completed — Lost to Follow-up | 22 | 17 | 0
Not completed — Non-Compliance with Study Drug | 4 | 1 | 0
Not completed — Physician Decision | 3 | 0 | 0
Not completed — Pregnancy | 8 | 8 | 0
Not completed — Withdrawal by Subject | 41 | 57 | 0
Not completed — No Longer Met Eligibility Criteria (for adolescents) | 14 | 29 | 0
Not completed — No Longer Met Eligibility Criteria (for adults) | 4 | 2 | 0
Not completed — Other | 10 | 4 | 0
Not completed — Approved Drug Available For Indication | 0 | 37 | 0
Period: Main Study: Treatment Period 2
Arm/Group | Main Study: Ritlecitinib 200 mg/ 50 mg QD (de Novo Participants) | Main Study: Ritlecitinib 50 mg QD (Roll-over Participants) | Vaccine Sub-study: Tdap With or Without Meningococcal ACWY Vaccine
Started | 289 | 332 | 0
Completed | 0 | 0 | 0
Not Completed | 289 | 332 | 0
Not completed — Adverse Event | 2 | 2 | 0
Not completed — Lack of Efficacy | 7 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 0
Not completed — Protocol Violation | 3 | 1 | 0
Not completed — Withdrawal by Subject | 8 | 7 | 0
Not completed — Other | 2 | 3 | 0
Not completed — Approved Drug Available For Indication | 179 | 222 | 0
Not completed — Ongoing | 86 | 96 | 0
Period: Main Study Observation Period
Arm/Group | Main Study: Ritlecitinib 200 mg/ 50 mg QD (de Novo Participants) | Main Study: Ritlecitinib 50 mg QD (Roll-over Participants) | Vaccine Sub-study: Tdap With or Without Meningococcal ACWY Vaccine
Started | 29 | 43 | 0
Completed | 1 | 1 | 0
Not Completed | 28 | 42 | 0
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Withdrawal by Subject | 10 | 14 | 0
Not completed — Other | 8 | 16 | 0
Not completed — Approved Drug Available For Indication | 6 | 9 | 0
Not completed — Ongoing | 2 | 1 | 0
Period: Vaccine Sub Study
Arm/Group | Main Study: Ritlecitinib 200 mg/ 50 mg QD (de Novo Participants) | Main Study: Ritlecitinib 50 mg QD (Roll-over Participants) | Vaccine Sub-study: Tdap With or Without Meningococcal ACWY Vaccine
Started | 0 | 0 | 17
Tdap Vaccination With or Without ACWY Vaccination | 0 | 0 | 17
ACWY Vaccination With Tdap Vaccination | 0 | 0 | 13
Completed (Participants who completed the 1-Month follow up visit of the vaccine sub-study) | 0 | 0 | 16
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis set comprised of all participants regardless of whether they received study intervention. Participants of main study and vaccine sub-study were not exclusive.
Groups:
- Total: Total of all reporting groups
Arm/Group | Main Study: Ritlecitinib 200 mg/ 50 mg QD (de Novo Participants) | Main Study: Ritlecitinib 50 mg QD (Roll-over Participants) | Vaccine Sub-study: Tdap With or Without Meningococcal ACWY Vaccine | Total
Number analyzed (Participants) | 449 | 603 | 17 | 1069
Age, Customized [Count of Participants; unit: Participants] — Population: Number Analyzed = number of participants analyzed for reporting arms of specified rows. Participants of main study and vaccine sub-study were not exclusive.
  Participants
    Main Study: number analyzed (Participants) | 449 | 603 | 0 | 1052
    Main Study: From 12 to <18 Years | 76 | 80 |  | 156
    Main Study: From 18 to <45 Years | 271 | 360 |  | 631
    Main Study: From 45 to <64 Years | 96 | 144 |  | 240
    Main Study: >=65 Years | 6 | 19 |  | 25
    Vaccine Substudy: number analyzed (Participants) | 0 | 0 | 17 | 17
    Vaccine Substudy: From 12 to <18 Years |  |  | 0 | 0
    Vaccine Substudy: From 18 to <45 Years |  |  | 10 | 10
    Vaccine Substudy: From 45 to <64 Years |  |  | 7 | 7
    Vaccine Substudy: >=65 Years |  |  | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Number Analyzed = number of participants analyzed for reporting arms of specified rows. Participants of main study and vaccine sub-study were not exclusive.
  Participants
    Main Study: number analyzed (Participants) | 449 | 603 | 0 | 1052
    Main Study: Female | 289 | 375 |  | 664
    Main Study: Male | 160 | 228 |  | 388
    Vaccine Substudy: number analyzed (Participants) | 0 | 0 | 17 | 17
    Vaccine Substudy: Female |  |  | 12 | 12
    Vaccine Substudy: Male |  |  | 5 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Number Analyzed = number of participants analyzed for reporting arms of specified rows. Participants of main study and vaccine sub-study were not exclusive.
  Participants
    Main Study: number analyzed (Participants) | 449 | 603 | 0 | 1052
    Main Study: Hispanic or Latino | 55 | 76 |  | 131
    Main Study: Not Hispanic or Latino | 383 | 523 |  | 906
    Main Study: Unknown or Not Reported | 11 | 4 |  | 15
    Vaccine Substudy: number analyzed (Participants) | 0 | 0 | 17 | 17
    Vaccine Substudy: Hispanic or Latino |  |  | 4 | 4
    Vaccine Substudy: Not Hispanic or Latino |  |  | 13 | 13
    Vaccine Substudy: Unknown or Not Reported |  |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Number Analyzed = number of participants analyzed for reporting arms of specified rows. Participants of main study and vaccine sub-study were not exclusive.
  Participants
    Main Study: number analyzed (Participants) | 449 | 603 | 0 | 1052
    Main Study: American Indian or Alaska Native | 5 | 3 |  | 8
    Main Study: Asian | 96 | 146 |  | 242
    Main Study: Native Hawaiian or Other Pacific Islander | 2 | 1 |  | 3
    Main Study: Black or African American | 16 | 21 |  | 37
    Main Study: White | 310 | 423 |  | 733
    Main Study: More than one race | 7 | 6 |  | 13
    Main Study: Unknown or Not Reported | 13 | 3 |  | 16
    Vaccine Substudy: number analyzed (Participants) | 0 | 0 | 17 | 17
    Vaccine Substudy: American Indian or Alaska Native |  |  | 0 | 0
    Vaccine Substudy: Asian |  |  | 3 | 3
    Vaccine Substudy: Native Hawaiian or Other Pacific Islander |  |  | 0 | 0
    Vaccine Substudy: Black or African American |  |  | 1 | 1
    Vaccine Substudy: White |  |  | 13 | 13
    Vaccine Substudy: More than one race |  |  | 0 | 0
    Vaccine Substudy: Unknown or Not Reported |  |  | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Main Study: Number of Participants With Treatment Emergent Adverse Events (TEAEs) Until Follow-up Visit
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE was considered treatment emergent if the event had start date on or after the first dosing date of this study.
Time Frame: From start of study intervention (Day 1) until follow-up visit (4 weeks after last dose in Treatment period 1) (Up to Month 40)
Population: SAS was defined as all participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Main Study: Ritlecitinib 200 mg/ 50 mg QD (de Novo Participants): Participants with a clinical diagnosis of AA received ritlecitinib (PF-06651600) 200 mg QD for 4 weeks followed by 50 mg ritlecitinib QD for 35 months during treatment period 1. After completion of treatment period 1, participants not continuing to treatment period 2 entered a follow-up period of 4 weeks. Participants from countries where ritlecitinib was not commercially available continued to receive 50 mg ritlecitinib QD in treatment period 2 for a maximum of 24 months or until availability of commercial product in their country, or until the sponsor terminated the study in that country, whichever occurred first. Participants who permanently discontinued study treatment entered an Observation Period where they completed the scheduled study visits for approximately 2 years or until study end, whichever occurred first.
Arm/Group | Main Study: Ritlecitinib 200 mg/ 50 mg QD (de Novo Participants) | Main Study: Ritlecitinib 50 mg QD (Roll-over Participants)
Number analyzed (Participants) | 447 | 603
Participants | 401 | 515

2. Primary Outcome: Main Study: Number of Participants With Serious Adverse Events (SAEs) and Adverse Events (AEs) Leading to Discontinuation Until Follow-up Visit
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An SAE was any untoward medical occurrence that at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life-threatening; resulted in persistent disability/incapacity; was a congenital anomaly/birth defect; other important medical events. AEs leading to discontinuation included participants who had an AE record that indicated that the AE caused the participant to be discontinued from the study or that action taken with study treatment was drug withdrawn.
Time Frame: as for outcome 1
Population: SAS was defined as all participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Ritlecitinib 200 mg/ 50 mg QD (de Novo Participants) | Main Study: Ritlecitinib 50 mg QD (Roll-over Participants)
Number analyzed (Participants) | 447 | 603
Participants
  SAEs | 30 | 42
  AEs Leading to Discontinuation | 36 | 46

3. Primary Outcome: Main Study: Number of Participants According to Categorization of Vital Signs Data Until Follow-up Visit
Description: Vital signs including blood pressure included systolic blood pressure (SBP) [Millimeters of mercury, mmHg]) and diastolic blood pressure (DBP) and pulse rate [beats per minute (bpm)] were measured using an automated device in a sitting position after at least 5 minutes of rest for the participant in a quiet setting without distractions. Criteria for vital sign abnormalities included: SBP<90mmHg, DBP<50 mmHg and pulse rate<40mmHg.
Time Frame: as for outcome 1
Population: SAS was defined as all participants who took at least 1 dose of study intervention. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Ritlecitinib 200 mg/ 50 mg QD (de Novo Participants) | Main Study: Ritlecitinib 50 mg QD (Roll-over Participants)
Number analyzed (Participants) | 443 | 600
Participants
  Diastolic blood pressure (mmHg): value <50 | 11 | 15
  Diastolic blood pressure (mmHg): change >=20 increase | 39 | 70
  Diastolic blood pressure (mmHg): change >=20 decrease | 45 | 51
  Pulse rate (bpm): Value <40 | 1 | 3
  Pulse rate (bpm): Value >120 | 0 | 1
  Systolic blood pressure (mmHg): Value <90 | 13 | 30
  Systolic blood pressure (mmHg): change>=30 increase | 18 | 42
  Systolic blood pressure (mmHg): change>=30 decrease | 22 | 30

4. Primary Outcome: Main Study: Number of Participants With Clinically Significant Abnormalities in Clinical Laboratory Values Until Follow-up Visit
Description: Criteria for laboratory abnormalities included:Hemoglobin, Hematocrit, Erythrocytes (<0.8*LLN); Ery. Volume, Hemoglobin,Mean Corpuscular HGB Concentration <0.8*LLN or >1.5*LLN;Reticulocytes, Leukocytes, Lymphocytes, Neutrophils, Neutrophils, Basophils, Eosinophils, Monocytes (>1.2*ULN), Prothrombin Time(>1.1*ULN).Clinical Chemistry: Bilirubin, Direct Bilirubin, Indirect Bilirubin (1.5*ULN), Aspartate Aminotransferase, Alanine Aminotransferase, Gamma Glutamyl Transferase, Alkaline Phosphatase (>3.0*ULN); Albumin, Urate (<0.8*LLN and >1.2*ULN; Urea Nitrogen,Creatinine Cholesterol >1.3*ULN; Cholesterol <0.8*LLN or >1.2*LLN, Triglycerides,Potassium,Calcium < 0.9x LLN & > 1.1x ULN; Bicarbonate, Glucose, Creatine Kinase. Urinalysis: Glucose, Ketones, Protein, Hemoglobin, Urobilinogen, Bilirubin, Nitrite >=1; Leukocyte Erythrocytes, Leukocytes >=20; Epithelial Cells>=6, Hyaline Cast>1; Bacteria>20. Number of participants with any laboratory abnormality meeting specified criteria is included.
Time Frame: as for outcome 1
Population: SAS was defined as all participants who took at least 1 dose of study intervention. Here, the "Overall number of participants analyzed" signifies the total number of participants evaluable for laboratory abnormalities, i.e. the number with at least one observation of the given laboratory test while on study treatment or during lag time (35 days after the last dose).
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Ritlecitinib 200 mg/ 50 mg QD (de Novo Participants) | Main Study: Ritlecitinib 50 mg QD (Roll-over Participants)
Number analyzed (Participants) | 444 | 602
Participants | 390 | 490

5. Primary Outcome: Vaccine Sub-study: Percentage of Participants With Tetanus Booster Response
Description: Booster response to tetanus toxoid was defined as: >=4-fold rise in anti-tetanus toxoid immunoglobulin G (IgG) antibody concentration at Month 1 if the pre-vaccination concentration was <=2.7 International Units per milliliter (IU/mL); OR >=2-fold rise in anti-tetanus toxoid IgG antibody concentration if the pre-vaccination concentration was >2.7 IU/mL. Two-sided 95% confidence interval (CI) was based on Clopper-Pearson exact method.
Time Frame: Month 1
Population: Safety Analysis Set (SAS) was defined as all participants from this sub-study who received at least 1 vaccine (Tdap or meningococcal ACWY). Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Vaccine Sub-study: Tdap Vaccination: Participants who have received atleast 6 months of treatment with PF-06651600 50mg QD in the study B7981032 were continued to receive the study intervention while participating in this vaccine sub-study. Eligible participants who received the Tdap vaccine with or without the meningococcal ACWY vaccine were enrolled in this sub-study.
Arm/Group | Vaccine Sub-study: Tdap Vaccination
Number analyzed (Participants) | 16
Percentage of participants | 62.5 [35.4 to 84.8]

6. Secondary Outcome: Main Study: Number of Participants With Treatment Emergent Adverse Events (TEAEs) Until End of Study
Description: as for outcome 1
Time Frame: From start of study intervention (Day 1) until end of study
Reporting Status: Not Posted, anticipated posting 2027-01

7. Secondary Outcome: Main Study: Number of Participants With Serious Adverse Events (SAEs) and Adverse Events (AEs) Leading to Discontinuation Until End of Study
Description: as for outcome 2
Time Frame: From start of study intervention (Day 1) until end of study
Reporting Status: Not Posted, anticipated posting 2027-01

8. Secondary Outcome: Main Study: Number of Participants With Clinically Significant Abnormalities in Vital Signs Until End of Study
Description: Vital signs including blood pressure (systolic and diastolic blood pressure [Millimeters of mercury, mmHg]) and pulse rate (beats per minute [bpm]) were measured using an automated device in a sitting position after at least 5 minutes of rest for the participant in a quiet setting without distractions. Clinically significant abnormalities will be determined by investigator.
Time Frame: From start of study intervention (Day 1) until end of study
Reporting Status: Not Posted, anticipated posting 2027-01

9. Secondary Outcome: Main Study: Number of Participants With Clinically Significant Laboratory Abnormalities Until End of Study
Description: Following laboratory parameters were assessed: Hemoglobin, Hematocrit, Erythrocytes Erythrocyte (ery.) corpuscular volume, Ery. Mean Corpuscular hemoglobin concentration, Reticulocytes, Leukocytes, Lymphocytes, Neutrophils, Basophils, Eosinophils, Monocytes, Prothrombin Time, Bilirubin, Direct Bilirubin, Indirect Bilirubin, Aspartate Aminotransferase, Alanine Aminotransferase, Gamma Glutamyl Transferase, Alkaline Phosphatase; Albumin, Urate; Urea Nitrogen, Creatinine, Cholesterol, Triglycerides, Potassium, Calcium, Bicarbonate, Glucose, Creatine Kinase. Urinalysis: Glucose, Ketones, Protein, Hemoglobin, Urobilinogen, Bilirubin, Nitrite, Leukocyte Erythrocytes, Leukocytes; Epithelial Cells, Hyaline Cast, Bacteria. Clinically significant abnormalities will be determined by investigator.
Time Frame: From start of study intervention (Day 1) until end of study
Reporting Status: Not Posted, anticipated posting 2027-01

10. Secondary Outcome: Main Study: Percentage of Participants Achieving Response Based on Severity of Alopecia Tool (SALT) Overall Score <=10 at Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 28, 32 and 36
Description: SALT is a quantitative assessment of AA severity based on the scalp terminal hair loss. A visual aid was utilized showing the division of the scalp hair into four quadrants (back, top of scalp, right side and left side), with each of the four quadrants given an accurate determination of the percentage of scalp surface area covered, representing 24%, 40%, 18%, and 18% of the total scalp surface area, respectively. Percentage of hair loss in these areas is multiplied by percent surface area of the scalp in that area. SALT score is the sum of percentage of hair loss in all areas and ranged from 0 (no hair loss) to 100 (complete scalp hair loss) with lower score indicating less hair loss. The SALT overall score included any hair loss regardless of etiology (e.g., including scalp hair loss due to both androgenetic alopecia and AA). In this outcome measure, percentage of participants with SALT overall score <= 10 were reported. 95% CI was calculated based on normal approximation.
Time Frame: At Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 28, 32 and 36
Population: Full Analysis Set (FAS) was defined as all participants regardless of whether they received study intervention. All participants reported under "Overall Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. Here, "Number Analyzed" signifies number of participants evaluable at specified time points.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Main Study: Ritlecitinib 200 mg/ 50 mg QD (de Novo Participants) | Main Study: Ritlecitinib 50 mg QD (Roll-over Participants)
Number analyzed (Participants) | 449 | 603
Percentage of participants
  Month 1: number analyzed (Participants) | 438 | 585
  Month 1 | 0.9 [0.02 to 1.80] | 27.9 [24.23 to 31.50]
  Month 3: number analyzed (Participants) | 423 | 580
  Month 3 | 16.3 [12.79 to 19.83] | 32.6 [28.77 to 36.40]
  Month 6: number analyzed (Participants) | 419 | 542
  Month 6 | 37.7 [33.07 to 42.35] | 39.1 [35.01 to 43.22]
  Month 9: number analyzed (Participants) | 398 | 510
  Month 9 | 49.0 [44.08 to 53.91] | 44.7 [40.39 to 49.02]
  Month 12: number analyzed (Participants) | 385 | 475
  Month 12 | 55.8 [50.88 to 60.80] | 48.2 [43.72 to 52.70]
  Month 15: number analyzed (Participants) | 368 | 448
  Month 15 | 59.5 [54.50 to 64.53] | 52.9 [48.28 to 57.52]
  Month 18: number analyzed (Participants) | 358 | 436
  Month 18 | 62.3 [57.27 to 67.31] | 53.4 [48.76 to 58.12]
  Month 21: number analyzed (Participants) | 345 | 430
  Month 21 | 62.9 [57.80 to 68.00] | 54.9 [50.18 to 59.59]
  Month 24: number analyzed (Participants) | 336 | 420
  Month 24 | 66.4 [61.32 to 71.42] | 56.4 [51.69 to 61.17]
  Month 28: number analyzed (Participants) | 319 | 410
  Month 28 | 68.3 [63.23 to 73.44] | 59.3 [54.51 to 64.02]
  Month 32: number analyzed (Participants) | 309 | 397
  Month 32 | 69.9 [64.79 to 75.02] | 61.0 [56.16 to 65.76]
  Month 36: number analyzed (Participants) | 296 | 373
  Month 36 | 70.9 [65.77 to 76.12] | 61.7 [56.73 to 66.60]

11. Secondary Outcome: Main Study: Percentage of Participants Achieving Response Based on Alopecia Areata (AA) SALT Score <=10 at Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 28, 32 and 36
Description: SALT is a quantitative assessment of AA severity based on scalp terminal hair loss. Scalp hair was divided into four quadrants (back, top of scalp, right side and left side), with each given an accurate determination of the percentage of scalp surface area covered, representing 24%, 40%, 18%, and 18% of the total scalp surface area, respectively. Percentage of hair loss in these areas is multiplied by percent surface area of scalp in that area. SALT score=sum of percentage of hair loss in all areas and ranged from 0 (no hair loss) to 100 (complete scalp hair loss) with lower score indicating less hair loss. SALT AA Score = SALT overall score minus SALT AGA score, where SALT overall score included any hair loss regardless of etiology and SALT AGA score included scalp hair loss only due to androgenetic alopecia. SALT AA score ranged from 0 (no hair loss) to 100 (complete scalp hair loss), with lower score indicating less hair loss. 95% CI was calculated based on normal approximation.
Time Frame: At Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 28, 32 and 36
Population: FAS was defined as all participants regardless of whether they received study intervention. All participants reported under "Overall Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. Here, "Overall Number Analyzed" signifies number of participants evaluable at specified time points.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Main Study: Ritlecitinib 200 mg/ 50 mg QD (de Novo Participants) | Main Study: Ritlecitinib 50 mg QD (Roll-over Participants)
Number analyzed (Participants) | 449 | 603
Percentage of participants
  Month 1: number analyzed (Participants) | 392 | 533
  Month 1 | 1.0 [0.03 to 2.02] | 28.5 [24.68 to 32.35]
  Month 3: number analyzed (Participants) | 378 | 534
  Month 3 | 17.7 [13.88 to 21.57] | 33.5 [29.52 to 37.52]
  Month 6: number analyzed (Participants) | 371 | 510
  Month 6 | 39.6 [34.65 to 44.60] | 39.8 [35.56 to 44.05]
  Month 9: number analyzed (Participants) | 359 | 483
  Month 9 | 50.7 [45.52 to 55.87] | 45.3 [40.90 to 49.78]
  Month 12: number analyzed (Participants) | 347 | 454
  Month 12 | 56.8 [51.56 to 61.98] | 49.3 [44.74 to 53.94]
  Month 15: number analyzed (Participants) | 334 | 432
  Month 15 | 61.4 [56.16 to 66.60] | 53.9 [49.23 to 58.64]
  Month 18: number analyzed (Participants) | 331 | 425
  Month 18 | 65.0 [59.81 to 70.09] | 54.1 [49.38 to 58.86]
  Month 21: number analyzed (Participants) | 325 | 419
  Month 21 | 65.2 [60.05 to 70.41] | 55.1 [50.37 to 59.89]
  Month 24: number analyzed (Participants) | 318 | 411
  Month 24 | 67.6 [62.47 to 72.75] | 57.2 [52.39 to 61.96]
  Month 28: number analyzed (Participants) | 305 | 403
  Month 28 | 69.2 [64.00 to 74.36] | 59.6 [54.76 to 64.35]
  Month 32: number analyzed (Participants) | 300 | 391
  Month 32 | 70.3 [65.16 to 75.50] | 61.6 [56.82 to 66.46]
  Month 36: number analyzed (Participants) | 294 | 372
  Month 36 | 71.1 [65.91 to 76.27] | 62.1 [57.17 to 67.03]

12. Secondary Outcome: Main Study: Percentage of Participants Achieving Response Based on SALT Overall Score <= 20 at Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 28, 32 and 36
Description: SALT is a quantitative assessment of AA severity based on the scalp terminal hair loss. A visual aid was utilized showing the division of the scalp hair into four quadrants (back, top of scalp, right side and left side), with each of the four quadrants given an accurate determination of the percentage of scalp surface area covered, representing 24%, 40%, 18%, and 18% of the total scalp surface area, respectively. Percentage of hair loss in these areas is multiplied by percent surface area of the scalp in that area. SALT score is the sum of percentage of hair loss in all areas and ranged from 0 (no hair loss) to 100 (complete scalp hair loss) with lower score indicating less hair loss. The SALT overall score included any hair loss regardless of etiology (e.g., including scalp hair loss due to both androgenetic alopecia and AA). In this outcome measure, percentage of participants with SALT overall score <=20 were reported. 95% CI was calculated based on normal approximation.
Time Frame: At Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 28, 32 and 36
Population: FAS was defined as all participants regardless of whether they received study intervention. All participants reported under "Overall Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. Here, "Number Analyzed" signifies number of participants evaluable at specified time points.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Main Study: Ritlecitinib 200 mg/ 50 mg QD (de Novo Participants) | Main Study: Ritlecitinib 50 mg QD (Roll-over Participants)
Number analyzed (Participants) | 449 | 603
Percentage of Participants
  Month 1: number analyzed (Participants) | 438 | 585
  Month 1 | 2.5 [1.05 to 3.98] | 35.6 [31.68 to 39.43]
  Month 3: number analyzed (Participants) | 423 | 580
  Month 3 | 27.7 [23.40 to 31.92] | 40.2 [36.18 to 44.16]
  Month 6: number analyzed (Participants) | 419 | 542
  Month 6 | 50.1 [45.33 to 54.91] | 50.4 [46.16 to 54.58]
  Month 9: number analyzed (Participants) | 398 | 510
  Month 9 | 59.5 [54.73 to 64.37] | 55.9 [51.57 to 60.19]
  Month 12: number analyzed (Participants) | 385 | 475
  Month 12 | 65.5 [60.70 to 70.20] | 60.0 [55.59 to 64.41]
  Month 15: number analyzed (Participants) | 368 | 448
  Month 15 | 70.7 [66.00 to 75.30] | 62.3 [57.79 to 66.77]
  Month 18: number analyzed (Participants) | 358 | 436
  Month 18 | 71.8 [67.13 to 76.45] | 63.5 [59.01 to 68.05]
  Month 21: number analyzed (Participants) | 345 | 430
  Month 21 | 72.8 [68.06 to 77.45] | 66.3 [61.81 to 70.75]
  Month 24: number analyzed (Participants) | 336 | 420
  Month 24 | 73.5 [68.79 to 78.23] | 66.7 [62.16 to 71.18]
  Month 28: number analyzed (Participants) | 319 | 410
  Month 28 | 76.8 [72.17 to 81.43] | 69.0 [64.55 to 73.50]
  Month 32: number analyzed (Participants) | 309 | 397
  Month 32 | 78.0 [73.37 to 82.61] | 69.5 [64.99 to 74.05]
  Month 36: number analyzed (Participants) | 296 | 373
  Month 36 | 79.1 [74.42 to 83.69] | 69.7 [65.04 to 74.37]

13. Secondary Outcome: Main Study: Percentage of Participants Achieving Response Based on AA SALT Score <=20 at Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 28, 32 and 36
Description: as for outcome 11
Time Frame: At Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 28, 32 and 36
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Main Study: Ritlecitinib 200 mg/ 50 mg QD (de Novo Participants) | Main Study: Ritlecitinib 50 mg QD (Roll-over Participants)
Number analyzed (Participants) | 449 | 603
Percentage of Participants
  Month 1: number analyzed (Participants) | 392 | 533
  Month 1 | 2.6 [0.99 to 4.11] | 36.6 [32.50 to 40.67]
  Month 3: number analyzed (Participants) | 378 | 534
  Month 3 | 27.8 [23.26 to 32.29] | 41.2 [37.02 to 45.37]
  Month 6: number analyzed (Participants) | 371 | 510
  Month 6 | 51.2 [46.13 to 56.30] | 51.0 [46.64 to 55.32]
  Month 9: number analyzed (Participants) | 359 | 483
  Month 9 | 60.4 [55.39 to 65.50] | 56.5 [52.10 to 60.94]
  Month 12: number analyzed (Participants) | 347 | 454
  Month 12 | 66.0 [61.01 to 70.98] | 61.2 [56.75 to 65.72]
  Month 15: number analyzed (Participants) | 334 | 432
  Month 15 | 72.2 [67.35 to 76.96] | 63.4 [58.88 to 67.97]
  Month 18: number analyzed (Participants) | 331 | 425
  Month 18 | 74.0 [69.29 to 78.74] | 64.5 [59.92 to 69.02]
  Month 21: number analyzed (Participants) | 325 | 419
  Month 21 | 74.2 [69.39 to 78.91] | 66.6 [62.07 to 71.10]
  Month 24: number analyzed (Participants) | 318 | 411
  Month 24 | 74.8 [70.07 to 79.61] | 66.9 [62.36 to 71.46]
  Month 28: number analyzed (Participants) | 305 | 403
  Month 28 | 77.7 [73.03 to 82.38] | 69.2 [64.72 to 73.74]
  Month 32: number analyzed (Participants) | 300 | 391
  Month 32 | 78.7 [74.03 to 83.30] | 69.3 [64.74 to 73.88]
  Month 36: number analyzed (Participants) | 294 | 372
  Month 36 | 79.3 [74.62 to 83.89] | 69.9 [65.23 to 74.55]

14. Secondary Outcome: Main Study: Change From Baseline in SALT Overall Score at Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 28, 32 and 36
Description: SALT is a quantitative assessment of AA severity based on the scalp terminal hair loss. A visual aid was utilized showing division of scalp hair into four quadrants (back, top of scalp, right side and left side), with each of four quadrants given an accurate determination of the percentage of scalp surface area covered, representing 24%, 40%, 18%, and 18% of total scalp surface area, respectively. Percentage of hair loss in these areas is multiplied by percent surface area of scalp in that area. SALT score is sum of percentage of hair loss in all areas and ranged from 0 (no hair loss) to 100 (complete scalp hair loss) with lower score indicating less hair loss. SALT overall score included any hair loss regardless of etiology (e.g., including scalp hair loss due to both androgenetic alopecia and AA). For roll-over participants originating from Study B7931005 or B7981015, baseline is day 1 from Study B7931005 or B7981015. For de novo participants, baseline is day 1 from Study B7981032.
Time Frame: Baseline, At Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 28, 32 and 36
Population: FAS was defined as all participants regardless of whether they received study intervention. Here, "Number Analyzed" signifies number of participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Main Study: Ritlecitinib 200 mg/ 50 mg QD (de Novo Participants) | Main Study: Ritlecitinib 50 mg QD (Roll-over Participants)
Number analyzed (Participants) | 449 | 603
Units on a scale
  Month 1: number analyzed (Participants) | 438 | 585
  Month 1 | -2.8 (9.94) | -41.8 (37.34)
  Month 3: number analyzed (Participants) | 423 | 580
  Month 3 | -23.6 (26.51) | -46.0 (37.32)
  Month 6: number analyzed (Participants) | 419 | 542
  Month 6 | -36.6 (32.07) | -52.0 (37.26)
  Month 9: number analyzed (Participants) | 398 | 510
  Month 9 | -44.2 (32.71) | -56.8 (35.89)
  Month 12: number analyzed (Participants) | 385 | 475
  Month 12 | -47.5 (32.34) | -60.1 (35.17)
  Month 15: number analyzed (Participants) | 368 | 448
  Month 15 | -50.6 (31.89) | -62.8 (33.88)
  Month 18: number analyzed (Participants) | 358 | 436
  Month 18 | -52.5 (31.98) | -64.2 (33.64)
  Month 21: number analyzed (Participants) | 345 | 430
  Month 21 | -53.3 (31.70) | -65.8 (32.43)
  Month 24: number analyzed (Participants) | 336 | 420
  Month 24 | -53.6 (31.79) | -65.5 (32.67)
  Month 28: number analyzed (Participants) | 319 | 410
  Month 28 | -54.8 (31.81) | -67.2 (32.49)
  Month 32: number analyzed (Participants) | 309 | 397
  Month 32 | -55.8 (31.48) | -67.8 (32.42)
  Month 36: number analyzed (Participants) | 296 | 373
  Month 36 | -56.6 (31.99) | -68.1 (32.17)

15. Secondary Outcome: Main Study: Change From Baseline in AA SALT Score at Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 28, 32 and 36
Description: SALT=quantitative assessment of AA severity based on scalp terminal hair loss. Scalp hair was divided into 4 quadrants (back, top of scalp, right side and left side), with each given an accurate determination of percentage of scalp surface area covered, representing 24%, 40%, 18%, and 18% of the total scalp surface area, respectively. Percentage of hair loss in these areas is multiplied by percent surface area of scalp in that area. SALT score=sum of percentage of hair loss in all areas and ranged from 0 (no hair loss) to 100 (complete scalp hair loss). SALT AA Score = SALT overall score minus SALT AGA score, where SALT overall score included any hair loss regardless of etiology and SALT AGA score included scalp hair loss only due to androgenetic alopecia. SALT AA score ranged from 0 (no hair loss) to 100 (complete scalp hair loss), lower score= less hair loss. Baseline (Roll-over participants: Day 1 from Study B7931005 or B7981015; De novo participants: Day 1 from Study B7981032).
Time Frame: Baseline, At Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 28, 32 and 36
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Main Study: Ritlecitinib 200 mg/ 50 mg QD (de Novo Participants) | Main Study: Ritlecitinib 50 mg QD (Roll-over Participants)
Number analyzed (Participants) | 449 | 603
Units on a scale
  Month 1: number analyzed (Participants) | 392 | 533
  Month 1 | -2.9 (10.32) | -42.8 (37.48)
  Month 3: number analyzed (Participants) | 378 | 534
  Month 3 | -23.8 (26.88) | -47.0 (37.33)
  Month 6: number analyzed (Participants) | 371 | 510
  Month 6 | -37.3 (32.12) | -52.8 (37.05)
  Month 9: number analyzed (Participants) | 359 | 483
  Month 9 | -44.8 (32.73) | -57.4 (35.81)
  Month 12: number analyzed (Participants) | 347 | 454
  Month 12 | -48.5 (32.20) | -61.1 (34.82)
  Month 15: number analyzed (Participants) | 334 | 432
  Month 15 | -51.6 (31.43) | -63.8 (33.41)
  Month 18: number analyzed (Participants) | 331 | 425
  Month 18 | -53.5 (31.39) | -65.0 (33.16)
  Month 21: number analyzed (Participants) | 325 | 419
  Month 21 | -53.8 (31.57) | -66.0 (32.43)
  Month 24: number analyzed (Participants) | 318 | 411
  Month 24 | -54.1 (31.93) | -65.9 (32.62)
  Month 28: number analyzed (Participants) | 305 | 403
  Month 28 | -55.2 (32.01) | -67.4 (32.53)
  Month 32: number analyzed (Participants) | 300 | 391
  Month 32 | -56.0 (31.69) | -67.8 (32.55)
  Month 36: number analyzed (Participants) | 294 | 371
  Month 36 | -56.5 (32.04) | -68.2 (32.18)

16. Secondary Outcome: Main Study: Percentage of Participants Achieving Atleast 75% Improvement in Overall SALT Score From Baseline at Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 28, 32 and 36
Description: SALT is a quantitative assessment of AA severity based on the scalp terminal hair loss. A visual aid was utilized showing the division of the scalp hair into four quadrants (back, top of scalp, right side and left side), with each of the four quadrants given an accurate determination of the percentage of scalp surface area covered, representing 24%, 40%, 18%, and 18% of the total scalp surface area, respectively. Percentage of hair loss in these areas is multiplied by percent surface area of the scalp in that area. SALT score is the sum of percentage of hair loss in all areas and ranged from 0 (no hair loss) to 100 (complete scalp hair loss) with lower score indicating less hair loss. The SALT overall score included any hair loss regardless of etiology (e.g., including scalp hair loss due to both androgenetic alopecia and AA). An Overall SALT 75 response was a 75% or greater reduction from baseline in SALT score.
Time Frame: At Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 28, 32 and 36
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Main Study: Ritlecitinib 200 mg/ 50 mg QD (de Novo Participants) | Main Study: Ritlecitinib 50 mg QD (Roll-over Participants)
Number analyzed (Participants) | 449 | 603
Percentage of participants
  Month 1: number analyzed (Participants) | 438 | 585
  Month 1 | 0.9 [0.02 to 1.80] | 37.4 [33.51 to 41.36]
  Month 3: number analyzed (Participants) | 423 | 580
  Month 3 | 21.5 [17.60 to 25.43] | 42.6 [38.56 to 46.61]
  Month 6: number analyzed (Participants) | 419 | 542
  Month 6 | 44.2 [39.40 to 48.91] | 51.3 [47.08 to 55.50]
  Month 9: number analyzed (Participants) | 398 | 510
  Month 9 | 55.5 [50.65 to 60.41] | 56.9 [52.56 to 61.16]
  Month 12: number analyzed (Participants) | 385 | 475
  Month 12 | 61.8 [56.97 to 66.67] | 61.3 [56.88 to 65.64]
  Month 15: number analyzed (Participants) | 368 | 448
  Month 15 | 67.4 [62.60 to 72.18] | 64.7 [60.31 to 69.16]
  Month 18: number analyzed (Participants) | 358 | 436
  Month 18 | 68.4 [63.62 to 73.25] | 66.7 [62.32 to 71.17]
  Month 21: number analyzed (Participants) | 345 | 430
  Month 21 | 69.3 [64.41 to 74.14] | 67.9 [63.49 to 72.32]
  Month 24: number analyzed (Participants) | 336 | 420
  Month 24 | 69.9 [65.04 to 74.84] | 68.1 [63.64 to 72.55]
  Month 28: number analyzed (Participants) | 319 | 410
  Month 28 | 73.4 [68.50 to 78.21] | 70.2 [65.82 to 74.67]
  Month 32: number analyzed (Participants) | 309 | 397
  Month 32 | 76.4 [71.64 to 81.11] | 70.5 [66.04 to 75.01]
  Month 36: number analyzed (Participants) | 296 | 373
  Month 36 | 76.7 [71.87 to 81.51] | 70.8 [66.16 to 75.39]

17. Secondary Outcome: Main Study: Percentage of Participants Achieving Atleast 75% Improvement in AA SALT Score From Baseline at Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 28, 32 and 36
Description: SALT=quantitative assessment of AA severity based on scalp terminal hair loss. Scalp hair was divided into four quadrants (back, top of scalp, right side and left side), with each given an accurate determination of percentage of scalp surface area covered, representing 24%, 40%, 18%, and 18% of the total scalp surface area, respectively. Percentage of hair loss in these areas is multiplied by percent surface area of scalp in that area. SALT score=sum of percentage of hair loss in all areas and ranged from 0 (no hair loss) to 100 (complete scalp hair loss) with lower score indicating less hair loss. SALT AA Score= SALT overall score minus SALT AGA score, where SALT overall score included any hair loss regardless of etiology and SALT AGA score included scalp hair loss only due to androgenetic alopecia. SALT AA score ranged from 0 (no hair loss) to 100 (complete scalp hair loss), where lower score=less hair loss. SALT 75 response= 75% or greater reduction from baseline in AA SALT score.
Time Frame: At Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 28, 32 and 36
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Main Study: Ritlecitinib 200 mg/ 50 mg QD (de Novo Participants) | Main Study: Ritlecitinib 50 mg QD (Roll-over Participants)
Number analyzed (Participants) | 449 | 603
Percentage of participants
  Month 1: number analyzed (Participants) | 392 | 533
  Month 1 | 1.0 [0.03 to 2.02] | 38.6 [34.52 to 42.78]
  Month 3: number analyzed (Participants) | 378 | 534
  Month 3 | 22.8 [18.53 to 26.98] | 43.6 [39.43 to 47.84]
  Month 6: number analyzed (Participants) | 371 | 510
  Month 6 | 45.6 [40.48 to 50.62] | 51.8 [47.43 to 56.10]
  Month 9: number analyzed (Participants) | 359 | 483
  Month 9 | 57.1 [51.98 to 62.22] | 57.3 [52.94 to 61.76]
  Month 12: number analyzed (Participants) | 347 | 454
  Month 12 | 62.8 [57.74 to 67.91] | 62.3 [57.88 to 66.79]
  Month 15: number analyzed (Participants) | 334 | 432
  Month 15 | 69.2 [64.21 to 74.11] | 65.5 [61.03 to 69.99]
  Month 18: number analyzed (Participants) | 331 | 425
  Month 18 | 70.7 [65.79 to 75.60] | 67.5 [63.08 to 71.98]
  Month 21: number analyzed (Participants) | 325 | 419
  Month 21 | 70.8 [65.82 to 75.71] | 68.0 [63.55 to 72.48]
  Month 24: number analyzed (Participants) | 318 | 411
  Month 24 | 72.0 [67.08 to 76.95] | 68.4 [63.87 to 72.87]
  Month 28: number analyzed (Participants) | 305 | 403
  Month 28 | 74.8 [69.88 to 79.63] | 70.5 [66.02 to 74.93]
  Month 32: number analyzed (Participants) | 300 | 391
  Month 32 | 77.3 [72.60 to 82.07] | 70.3 [65.80 to 74.86]
  Month 36: number analyzed (Participants) | 294 | 371
  Month 36 | 77.2 [72.42 to 82.01] | 70.9 [66.27 to 75.51]

18. Secondary Outcome: Main Study: Percentage of Participants Achieving Atleast 2-Grade Improvement From Baseline or Absolute Score of 3 in the Eyebrow Assessment (EBA) at Months 1, 3, 6, 12, 18, 24 and 36 in Participants Without Normal EBA Score at Baseline
Description: EBA is a numeric rating scale developed to characterize eyebrow hair loss. The numeric rating scale ranges from 0 (none) to 3 (normal), where 0= no eyebrow, 1=minimal eyebrow, 2=moderate eyebrow and 3= normal eyebrow. Higher scores represent lesser loss of eyebrow hair. 95% CI was based on normal approximation.
Time Frame: At Months 1, 3, 6, 12, 18, 24 and 36
Population: FAS was defined as all participants regardless of whether they received study intervention. All participants reported under "Number of Participants Analyzed" included all participants from FAS without normal EBA score at baseline who contributed data to the table; however, may not have evaluable data for every row. Here, "Number Analyzed" signifies number of participants evaluable at specified time points.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Main Study: Ritlecitinib 200 mg/ 50 mg QD (de Novo Participants) | Main Study: Ritlecitinib 50 mg QD (Roll-over Participants)
Number analyzed (Participants) | 449 | 603
Percentage of participants
  Month 1: number analyzed (Participants) | 324 | 482
  Month 1 | 4.3 [2.11 to 6.53] | 38.8 [34.45 to 43.15]
  Month 3: number analyzed (Participants) | 314 | 475
  Month 3 | 22.3 [17.69 to 26.90] | 43.4 [38.91 to 47.83]
  Month 6: number analyzed (Participants) | 311 | 446
  Month 6 | 37.6 [32.24 to 43.00] | 50.0 [45.36 to 54.64]
  Month 12: number analyzed (Participants) | 280 | 388
  Month 12 | 55.0 [49.17 to 60.83] | 60.3 [55.44 to 65.18]
  Month 18: number analyzed (Participants) | 264 | 358
  Month 18 | 59.5 [53.55 to 65.39] | 64.2 [59.28 to 69.21]
  Month 24: number analyzed (Participants) | 245 | 343
  Month 24 | 61.2 [55.12 to 67.33] | 67.9 [62.99 to 72.87]
  Month 36: number analyzed (Participants) | 215 | 309
  Month 36 | 65.6 [59.23 to 71.93] | 69.9 [64.79 to 75.02]

19. Secondary Outcome: Main Study: Percentage of Participants Achieving Atleast 2-Grade Improvement From Baseline or Absolute Score of 3 in the Eyelash Assessment (ELA) at Months 1, 3, 6, 12, 18, 24 and 36 in Participants Without Normal ELA Score at Baseline
Description: ELA is a numeric rating scale developed to characterize eyelash hair loss. The numeric rating scale ranges from 0 (none) to 3 (normal), where 0=no eyelash, 1=minimal eyelash, 2=moderate eyelash and 3=normal eyelash. Higher scores represent lesser loss of eyelash hair.
Time Frame: At Months 1, 3, 6, 12, 18, 24 and 36
Population: FAS was defined as all participants regardless of whether they received study intervention. All participants reported under "Overall Number of Participants Analyzed" included all participants from FAS without normal ELA score at baseline who contributed data to the table; however, may not have evaluable data for every row. Here, "Number Analyzed" signifies number of participants evaluable at specified time points.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Main Study: Ritlecitinib 200 mg/ 50 mg QD (de Novo Participants) | Main Study: Ritlecitinib 50 mg QD (Roll-over Participants)
Number analyzed (Participants) | 449 | 603
Percentage of participants
  Month 1: number analyzed (Participants) | 291 | 440
  Month 1 | 3.4 [1.34 to 5.53] | 37.7 [33.20 to 42.26]
  Month 3: number analyzed (Participants) | 282 | 435
  Month 3 | 17.7 [13.27 to 22.19] | 42.5 [37.88 to 47.17]
  Month 6: number analyzed (Participants) | 278 | 410
  Month 6 | 36.7 [31.03 to 42.36] | 47.1 [42.24 to 51.90]
  Month 12: number analyzed (Participants) | 250 | 354
  Month 12 | 54.8 [48.63 to 60.97] | 56.5 [51.33 to 61.66]
  Month 18: number analyzed (Participants) | 235 | 327
  Month 18 | 62.1 [55.93 to 68.33] | 61.2 [55.88 to 66.44]
  Month 24: number analyzed (Participants) | 216 | 313
  Month 24 | 66.2 [59.90 to 72.51] | 68.1 [62.89 to 73.22]
  Month 36: number analyzed (Participants) | 186 | 278
  Month 36 | 69.4 [62.73 to 75.98] | 70.5 [65.14 to 75.86]

20. Secondary Outcome: Main Study: Percentage of Participants Achieving Patient's Global Impression of Change (PGI-C) Score of Moderately Improved or Greatly Improved at Months 1, 3, 6, 9, 12, 18, 24 and 36
Description: PGI-C is a self-administered single item questionnaire to evaluate the improvement or worsening of participant's AA as compared to the start of the study. Participants were required to select their response on a 7-point scale ranging from 1 (greatly worsened), 2=moderately worsened, 3=slightly worsened, 4=not changed, 5= slightly improved, 6=moderately improved, 7 (greatly improved). 95% CI was based on normal approximation.
Time Frame: At Months 1, 3, 6, 9, 12, 18, 24 and 36
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Main Study: Ritlecitinib 200 mg/ 50 mg QD (de Novo Participants) | Main Study: Ritlecitinib 50 mg QD (Roll-over Participants)
Number analyzed (Participants) | 449 | 603
Percentage of participants
  Month 1: number analyzed (Participants) | 438 | 587
  Month 1 | 16.4 [12.97 to 19.91] | 55.2 [51.17 to 59.22]
  Month 3: number analyzed (Participants) | 426 | 580
  Month 3 | 57.0 [52.34 to 61.74] | 59.3 [55.31 to 63.31]
  Month 6: number analyzed (Participants) | 423 | 542
  Month 6 | 68.8 [64.38 to 73.21] | 66.4 [62.44 to 70.40]
  Month 9: number analyzed (Participants) | 396 | 509
  Month 9 | 76.5 [72.34 to 80.69] | 69.5 [65.55 to 73.55]
  Month 12: number analyzed (Participants) | 384 | 474
  Month 12 | 78.6 [74.55 to 82.74] | 72.6 [68.56 to 76.59]
  Month 18: number analyzed (Participants) | 357 | 436
  Month 18 | 81.0 [76.88 to 85.03] | 74.8 [70.69 to 78.85]
  Month 24: number analyzed (Participants) | 335 | 420
  Month 24 | 82.4 [78.31 to 86.47] | 78.6 [74.65 to 82.50]
  Month 36: number analyzed (Participants) | 295 | 372
  Month 36 | 83.1 [78.77 to 87.33] | 79.0 [74.90 to 83.17]

21. Secondary Outcome: Main Study: Change From Baseline in Alopecia Areata Patient Priority Outcomes (AAPPO) Domain Scores at Months 1, 3, 6, 9, 12, 18, 24 and 36: Emotional Symptoms and Activity Limitations
Description: AAPPO scale is a 11-item self-administered questionnaire that measured hair loss, emotional symptoms, and activity limitations over past week. Items 5-8 assessed emotional symptoms with responses scored from 0 ='never' to 4='always'. Items 9-11 assessed activity limitations with responses scored from 0='not at all' to 4='completely'. AAPPO emotional symptoms sub score was calculated as mean of items 5-8 and ranged from 0 (never) to 4 (always), where higher scores indicated more emotional symptoms. AAPPO activity limitations sub score was calculated as mean of items 9-11 and ranged from 0(not at all) to 4(completely), where higher scores indicated more activity limitations. For roll-over participants originating from Study B7931005 or B7981015, baseline is day 1 from Study B7931005 or B7981015. For de novo participants, baseline is day 1 from Study B7981032.
Time Frame: Baseline, At Months 1, 3, 6, 9, 12, 18, 24 and 36
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Main Study: Ritlecitinib 200 mg/ 50 mg QD (de Novo Participants) | Main Study: Ritlecitinib 50 mg QD (Roll-over Participants)
Number analyzed (Participants) | 449 | 603
Units on a scale
  Month 1: Emotional Symptoms: number analyzed (Participants) | 434 | 584
  Month 1: Emotional Symptoms | -0.33 (0.683) | -0.84 (1.036)
  Month 3: Emotional Symptoms: number analyzed (Participants) | 427 | 576
  Month 3: Emotional Symptoms | -0.61 (0.867) | -0.86 (1.055)
  Month 6: Emotional Symptoms: number analyzed (Participants) | 424 | 534
  Month 6: Emotional Symptoms | -0.77 (1.012) | -0.95 (1.087)
  Month 9: Emotional Symptoms: number analyzed (Participants) | 398 | 505
  Month 9: Emotional Symptoms | -0.95 (1.091) | -0.95 (1.123)
  Month 12: Emotional Symptoms: number analyzed (Participants) | 385 | 471
  Month 12: Emotional Symptoms | -1.00 (1.161) | -1.04 (1.128)
  Month 18: Emotional Symptoms: number analyzed (Participants) | 357 | 434
  Month 18: Emotional Symptoms | -1.07 (1.174) | -1.11 (1.129)
  Month 24: Emotional Symptoms: number analyzed (Participants) | 335 | 417
  Month 24: Emotional Symptoms | -1.12 (1.232) | -1.07 (1.172)
  Month 36: Emotional Symptoms: number analyzed (Participants) | 295 | 368
  Month 36: Emotional Symptoms | -1.20 (1.246) | -1.11 (1.204)
  Month 1: Activity Limitations: number analyzed (Participants) | 434 | 584
  Month 1: Activity Limitations | -0.09 (0.641) | -0.36 (0.789)
  Month 3: Activity Limitations: number analyzed (Participants) | 427 | 576
  Month 3: Activity Limitations | -0.21 (0.667) | -0.38 (0.811)
  Month 6: Activity Limitations: number analyzed (Participants) | 424 | 534
  Month 6: Activity Limitations | -0.27 (0.719) | -0.44 (0.829)
  Month 9: Activity Limitations: number analyzed (Participants) | 398 | 506
  Month 9: Activity Limitations | -0.33 (0.781) | -0.45 (0.857)
  Month 12: Activity Limitations: number analyzed (Participants) | 385 | 471
  Month 12: Activity Limitations | -0.36 (0.793) | -0.51 (0.871)
  Month 18: Activity Limitations: number analyzed (Participants) | 358 | 434
  Month 18: Activity Limitations | -0.40 (0.830) | -0.51 (0.869)
  Month 24: Activity Limitations: number analyzed (Participants) | 335 | 416
  Month 24: Activity Limitations | -0.43 (0.824) | -0.52 (0.890)
  Month 36: Activity Limitations: number analyzed (Participants) | 295 | 368
  Month 36: Activity Limitations | -0.43 (0.858) | -0.53 (0.859)

22. Secondary Outcome: Main Study: Percentage of Participants With Response Based on Hair Loss Improvement From Baseline in Alopecia Areata Patient Priority Outcomes (AAPPO) Domain Scores at Months 1, 3, 6, 9, 12, 18, 24 and 36, Among Participants With Score >=2 at Baseline
Description: AAPPO scale is a 11-item self-administered questionnaire that measured hair loss, emotional symptoms, and activity limitations over past week. Items 1-4 assessed current hair loss from the scalp, eyebrows, eyelashes and body using a 5 point scale that ranged from 0 ='no hair loss' and 4='complete hair loss'. In this outcome measure, percentage of participants with AAPPO domain scores of 0 = no hair loss or 1 = a little hair loss, among participants with score >=2 at baseline are reported.
Time Frame: Baseline, At Months 1, 3, 6, 9, 12, 18, 24 and 36
Population: FAS was defined as all participants regardless of whether they received study intervention. Participants reported under "Overall Number of Participants Analyzed" included all participants from FAS who had an AAPPO baseline score >=2 who contributed data to the table; however, may not have evaluable data for every row. Here, "Number Analyzed" signifies number of participants evaluable at specified time points.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Main Study: Ritlecitinib 200 mg/ 50 mg QD (de Novo Participants) | Main Study: Ritlecitinib 50 mg QD (Roll-over Participants)
Number analyzed (Participants) | 449 | 603
Percentage of participants
  Month 1: Current hair loss on Scalp: number analyzed (Participants) | 418 | 567
  Month 1: Current hair loss on Scalp | 9.8 [6.96 to 12.66] | 37.2 [33.23 to 41.19]
  Month 3: Current hair loss on Scalp: number analyzed (Participants) | 411 | 559
  Month 3: Current hair loss on Scalp | 27.5 [23.18 to 31.81] | 38.5 [34.43 to 42.49]
  Month 6: Current hair loss on Scalp: number analyzed (Participants) | 409 | 517
  Month 6: Current hair loss on Scalp | 45.7 [40.89 to 50.55] | 46.4 [42.12 to 50.72]
  Month 9: Current hair loss on Scalp: number analyzed (Participants) | 383 | 490
  Month 9: Current hair loss on Scalp | 55.6 [50.64 to 60.59] | 49.8 [45.37 to 54.22]
  Month 12: Current hair loss on Scalp: number analyzed (Participants) | 370 | 459
  Month 12: Current hair loss on Scalp | 58.9 [53.91 to 63.93] | 52.7 [48.16 to 57.29]
  Month 18: Current hair loss on Scalp: number analyzed (Participants) | 347 | 421
  Month 18: Current hair loss on Scalp | 62.2 [57.15 to 67.35] | 57.2 [52.52 to 61.97]
  Month 24: Current hair loss on Scalp: number analyzed (Participants) | 326 | 402
  Month 24: Current hair loss on Scalp | 67.8 [62.72 to 72.86] | 60.7 [55.92 to 65.47]
  Month 36: Current hair loss on Scalp: number analyzed (Participants) | 287 | 354
  Month 36: Current hair loss on Scalp | 69.3 [64.00 to 74.67] | 58.5 [53.34 to 63.61]
  Month 1: Current hair loss on Eyebrows: number analyzed (Participants) | 274 | 441
  Month 1: Current hair loss on Eyebrows | 9.9 [6.33 to 13.38] | 42.9 [38.24 to 47.48]
  Month 3: Current hair loss on Eyebrows: number analyzed (Participants) | 272 | 433
  Month 3: Current hair loss on Eyebrows | 32.4 [26.79 to 37.91] | 44.1 [39.43 to 48.79]
  Month 6: Current hair loss on Eyebrows: number analyzed (Participants) | 269 | 398
  Month 6: Current hair loss on Eyebrows | 43.9 [37.94 to 49.80] | 49.5 [44.59 to 54.41]
  Month 9: Current hair loss on Eyebrows: number analyzed (Participants) | 247 | 376
  Month 9: Current hair loss on Eyebrows | 49.0 [42.75 to 55.22] | 52.9 [47.88 to 57.97]
  Month 12: Current hair loss on Eyebrows: number analyzed (Participants) | 236 | 347
  Month 12: Current hair loss on Eyebrows | 55.5 [49.17 to 61.85] | 55.0 [49.81 to 60.28]
  Month 18: Current hair loss on Eyebrows: number analyzed (Participants) | 220 | 321
  Month 18: Current hair loss on Eyebrows | 60.9 [54.46 to 67.36] | 60.1 [54.77 to 65.48]
  Month 24: Current hair loss on Eyebrows: number analyzed (Participants) | 201 | 309
  Month 24: Current hair loss on Eyebrows | 60.7 [53.94 to 67.45] | 64.4 [59.06 to 69.74]
  Month 36: Current hair loss on Eyebrows: number analyzed (Participants) | 174 | 275
  Month 36: Current hair loss on Eyebrows | 63.8 [56.65 to 70.93] | 64.7 [59.08 to 70.37]
  Month 1: Current hair loss on Eyelashes: number analyzed (Participants) | 235 | 386
  Month 1: Current hair loss on Eyelashes | 8.1 [4.60 to 11.57] | 40.9 [36.03 to 45.84]
  Month 3: Current hair loss on Eyelashes: number analyzed (Participants) | 232 | 380
  Month 3: Current hair loss on Eyelashes | 35.8 [29.61 to 41.94] | 44.2 [39.22 to 49.20]
  Month 6: Current hair loss on Eyelashes: number analyzed (Participants) | 230 | 350
  Month 6: Current hair loss on Eyelashes | 45.7 [39.21 to 52.09] | 46.6 [41.35 to 51.80]
  Month 9: Current hair loss on Eyelashes: number analyzed (Participants) | 212 | 328
  Month 9: Current hair loss on Eyelashes | 54.2 [47.54 to 60.95] | 54.0 [48.57 to 59.36]
  Month 12: Current hair loss on Eyelashes: number analyzed (Participants) | 201 | 309
  Month 12: Current hair loss on Eyelashes | 56.2 [49.36 to 63.08] | 55.3 [49.80 to 60.88]
  Month 18: Current hair loss on Eyelashes: number analyzed (Participants) | 189 | 281
  Month 18: Current hair loss on Eyelashes | 61.9 [54.98 to 68.83] | 62.3 [56.61 to 67.94]
  Month 24: Current hair loss on Eyelashes: number analyzed (Participants) | 171 | 266
  Month 24: Current hair loss on Eyelashes | 64.3 [57.15 to 71.51] | 65.0 [59.31 to 70.77]
  Month 36: Current hair loss on Eyelashes: number analyzed (Participants) | 149 | 237
  Month 36: Current hair loss on Eyelashes | 69.8 [62.43 to 77.17] | 67.5 [61.55 to 73.47]
  Month 1: Current hair loss on body: number analyzed (Participants) | 279 | 436
  Month 1: Current hair loss on body | 14.7 [10.54 to 18.85] | 31.9 [27.51 to 36.25]
  Month 3: Current hair loss on body: number analyzed (Participants) | 276 | 430
  Month 3: Current hair loss on body | 24.3 [19.22 to 29.33] | 36.5 [31.96 to 41.06]
  Month 6: Current hair loss on body: number analyzed (Participants) | 272 | 396
  Month 6: Current hair loss on body | 34.6 [28.91 to 40.21] | 41.9 [37.06 to 46.78]
  Month 9: Current hair loss on body: number analyzed (Participants) | 252 | 371
  Month 9: Current hair loss on body | 43.7 [37.53 to 49.77] | 46.9 [41.82 to 51.98]
  Month 12: Current hair loss on body: number analyzed (Participants) | 243 | 347
  Month 12: Current hair loss on body | 52.3 [45.98 to 58.54] | 49.9 [44.60 to 55.12]
  Month 18: Current hair loss on body: number analyzed (Participants) | 227 | 318
  Month 18: Current hair loss on body | 55.9 [49.49 to 62.41] | 56.0 [50.52 to 61.43]
  Month 24: Current hair loss on body: number analyzed (Participants) | 208 | 302
  Month 24: Current hair loss on body | 59.1 [52.45 to 65.82] | 60.3 [54.75 to 65.78]
  Month 36: Current hair loss on body: number analyzed (Participants) | 181 | 270
  Month 36: Current hair loss on body | 65.2 [58.25 to 72.13] | 62.2 [56.44 to 68.01]

23. Secondary Outcome: Main Study: Change From Baseline in Depression Subscale Score of Hospital Anxiety and Depression Scale (HADS) at Months 1, 3, 6, 9, 12, 18, 24 and 36
Description: HADS is a validated 14-item questionnaire used to assess states of anxiety and depression over the past week. The HADS consisted of 2 subscales, one for anxiety (HADS-A) and one for depression (HADS-D). The depression subscale comprised of 7 items with score ranging from 0 (no presence of depression) to 3 (severe feeling of depression). Total depression subscale score was calculated as the sum of 7 items and ranged from 0 to 21; higher score indicating greater severity of depression symptoms. For roll-over participants originating from Study B7931005 or B7981015, baseline is day 1 from Study B7931005 or B7981015. For de novo participants, baseline is day 1 from Study B7981032.
Time Frame: Baseline, At Months 1, 3, 6, 9, 12, 18, 24 and 36
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Main Study: Ritlecitinib 200 mg/ 50 mg QD (de Novo Participants) | Main Study: Ritlecitinib 50 mg QD (Roll-over Participants)
Number analyzed (Participants) | 449 | 603
Units on a scale
  Month 1: number analyzed (Participants) | 431 | 587
  Month 1 | -0.1 (2.27) | -0.6 (2.87)
  Month 3: number analyzed (Participants) | 426 | 578
  Month 3 | -0.4 (2.47) | -0.5 (2.80)
  Month 6: number analyzed (Participants) | 422 | 540
  Month 6 | -0.5 (2.60) | -0.7 (2.97)
  Month 9: number analyzed (Participants) | 397 | 508
  Month 9 | -0.6 (2.64) | -0.9 (2.94)
  Month 12: number analyzed (Participants) | 385 | 471
  Month 12 | -0.6 (2.66) | -0.9 (3.16)
  Month 18: number analyzed (Participants) | 357 | 436
  Month 18 | -0.9 (2.72) | -0.9 (3.08)
  Month 24: number analyzed (Participants) | 335 | 420
  Month 24 | -1.0 (2.75) | -1.1 (3.11)
  Month 36: number analyzed (Participants) | 295 | 366
  Month 36 | -0.8 (2.92) | -1.0 (2.90)

24. Secondary Outcome: Main Study: Change From Baseline in Anxiety Subscale Score of Hospital Anxiety and Depression Scale (HADS) at Months 1, 3, 6, 9, 12, 18, 24 and 36
Description: HADS is a validated 14-item questionnaire used to assess states of anxiety and depression over the past week. The HADS consisted of 2 subscales, one for anxiety (HADS-A) and one for depression (HADS-D). The anxiety subscale comprised of 7 items with score ranging from 0 (no anxiety) to 3 (severe anxiety). Total anxiety subscale score was calculated as the sum of 7 items and ranged from 0 to 21; higher score indicating greater severity of anxiety symptoms. For roll-over participants originating from Study B7931005 or B7981015, baseline is day 1 from Study B7931005 or B7981015. For de novo participants, baseline is day 1 from Study B7981032.
Time Frame: Baseline, At Months 1, 3, 6, 9, 12, 18, 24 and 36
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Main Study: Ritlecitinib 200 mg/ 50 mg QD (de Novo Participants) | Main Study: Ritlecitinib 50 mg QD (Roll-over Participants)
Number analyzed (Participants) | 449 | 603
Units on a scale
  Month 1: number analyzed (Participants) | 430 | 586
  Month 1 | -0.6 (2.57) | -0.9 (3.38)
  Month 3: number analyzed (Participants) | 425 | 575
  Month 3 | -0.7 (2.65) | -0.9 (3.46)
  Month 6: number analyzed (Participants) | 420 | 539
  Month 6 | -0.9 (2.79) | -1.2 (3.33)
  Month 9: number analyzed (Participants) | 395 | 506
  Month 9 | -0.9 (3.02) | -1.1 (3.46)
  Month 12: number analyzed (Participants) | 384 | 471
  Month 12 | -0.8 (3.14) | -1.1 (3.52)
  Month 18: number analyzed (Participants) | 356 | 435
  Month 18 | -1.0 (3.01) | -1.1 (3.45)
  Month 24: number analyzed (Participants) | 334 | 419
  Month 24 | -1.1 (3.21) | -1.2 (3.48)
  Month 36: number analyzed (Participants) | 294 | 365
  Month 36 | -1.0 (3.35) | -1.1 (3.46)

25. Secondary Outcome: Main Study: Percentage of Participants With Improvement on HADS Depression Score at Months 1, 3, 6, 9, 12, 18, 24 and 36
Description: HADS is a validated 14-item questionnaire used to assess states of anxiety and depression over the past week. The HADS consisted of 2 subscales, one for anxiety (HADS-A) and one for depression (HADS-D). The depression subscale comprised of 7 items with score ranging from 0 (no presence of depression) to 3 (severe feeling of depression). Total depression subscale score was calculated as the sum of 7 items and ranged from 0 to 21; higher score indicating greater severity of depression symptoms. Improvement on HADS depression score was considered as achieving a "normal" depression subscale score indicative of an absence of depression. Among adults, a HADS-D score of 0-7 was considered "normal"; for adolescents, a HADS-D score of 0-6 was considered "normal". 95% CI was calculated based on normal approximation.
Time Frame: At Months 1, 3, 6, 9, 12, 18, 24 and 36
Population: FAS included was defined as all participants regardless of whether they received study intervention. All participants reported under "Overall Number of Participants Analyzed" included all participants from the FAS with a score indicative of depression at baseline who contributed data to the table; however, may not have evaluable data for every row. Here, "Number Analyzed" signifies number of participants evaluable at specified time points.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Main Study: Ritlecitinib 200 mg/ 50 mg QD (de Novo Participants) | Main Study: Ritlecitinib 50 mg QD (Roll-over Participants)
Number analyzed (Participants) | 36 | 59
Percentage of participants
  Month 1: number analyzed (Participants) | 32 | 58
  Month 1 | 53.1 [35.84 to 70.41] | 56.9 [44.15 to 69.64]
  Month 3: number analyzed (Participants) | 30 | 57
  Month 3 | 63.3 [46.09 to 80.58] | 52.6 [39.67 to 65.59]
  Month 6: number analyzed (Participants) | 30 | 54
  Month 6 | 70.0 [53.60 to 86.40] | 70.4 [58.19 to 82.55]
  Month 9: number analyzed (Participants) | 29 | 49
  Month 9 | 65.5 [48.22 to 82.82] | 69.4 [56.48 to 82.29]
  Month 12: number analyzed (Participants) | 29 | 44
  Month 12 | 58.6 [40.70 to 76.55] | 72.7 [59.57 to 85.89]
  Month 18: number analyzed (Participants) | 26 | 44
  Month 18 | 84.6 [70.75 to 98.48] | 63.6 [49.42 to 77.85]
  Month 24: number analyzed (Participants) | 24 | 43
  Month 24 | 83.3 [68.42 to 98.24] | 62.8 [48.34 to 77.24]
  Month 36: number analyzed (Participants) | 20 | 37
  Month 36 | 80.0 [62.47 to 97.53] | 75.7 [61.85 to 89.50]

26. Secondary Outcome: Main Study: Percentage of Participants With Improvement on HADS Anxiety Score At Months 1, 3, 6, 9, 12, 18, 24 and 36
Description: HADS is a validated 14-item questionnaire used to assess states of anxiety and depression over the past week. The HADS consisted of 2 subscales, one for anxiety (HADS-A) and one for depression (HADS-D). The anxiety subscale comprised of 7 items with score ranging from 0 (no anxiety) to 3 (severe anxiety). Total anxiety subscale score was calculated as the sum of 7 items and ranged from 0 to 21; higher score indicating greater severity of anxiety symptoms. Improvement on HADS anxiety score was considered as achieving a "normal" anxiety subscale score indicative of an absence of anxiety. Among adults, a HADS-A score of 0-7 was considered "normal"; for adolescents, a HADS-A score of 0-8 was considered "normal". 95% CI was calculated based on normal approximation.
Time Frame: At Months 1, 3, 6, 9, 12, 18, 24 and 36
Population: FAS was defined as all participants regardless of whether they received study intervention. All participants reported under "Overall Number of Participants Analyzed" included all participants from the FAS with a score indicative of anxiety at baseline who contributed data to the table; however, may not have evaluable data for every row. Here, "Number Analyzed" signifies number of participants evaluable at specified time points.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Main Study: Ritlecitinib 200 mg/ 50 mg QD (de Novo Participants) | Main Study: Ritlecitinib 50 mg QD (Roll-over Participants)
Number analyzed (Participants) | 95 | 122
Percentage of participants
  Month 1: number analyzed (Participants) | 88 | 118
  Month 1 | 51.1 [40.69 to 61.58] | 54.2 [45.25 to 63.23]
  Month 3: number analyzed (Participants) | 86 | 114
  Month 3 | 46.5 [35.97 to 57.05] | 59.6 [50.64 to 68.65]
  Month 6: number analyzed (Participants) | 84 | 112
  Month 6 | 53.6 [42.91 to 64.24] | 62.5 [53.53 to 71.47]
  Month 9: number analyzed (Participants) | 78 | 109
  Month 9 | 50.0 [38.90 to 61.10] | 57.8 [48.53 to 67.07]
  Month 12: number analyzed (Participants) | 79 | 104
  Month 12 | 54.4 [43.45 to 65.41] | 64.4 [55.22 to 73.62]
  Month 18: number analyzed (Participants) | 73 | 97
  Month 18 | 69.9 [59.34 to 80.39] | 62.9 [53.27 to 72.50]
  Month 24: number analyzed (Participants) | 67 | 95
  Month 24 | 73.1 [62.52 to 83.75] | 61.1 [51.25 to 70.86]
  Month 36: number analyzed (Participants) | 58 | 83
  Month 36 | 62.1 [49.58 to 74.56] | 63.9 [53.52 to 74.19]

27. Secondary Outcome: Vaccine Sub-study: Percentage of Participants With Anti-tetanus Antibody Level >=1.0 International Units Per Milliliter (IU/mL) at Month 1-Tdap Vaccination
Description: Percentage of participants with anti-tetanus antibody level >=1.0 IU/mL at Month 1 were reported in this outcome measure. Two-sided 95% CI was based on Clopper-Pearson exact method.
Time Frame: Month 1
Population: FAS-Tdap was defined as all participants who received the Tdap vaccine (with or without the meningococcal ACWY vaccine). Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Vaccine Sub-study: Tdap Vaccination
Number analyzed (Participants) | 16
Percentage of participants | 100 [79.4 to 100.0]

28. Secondary Outcome: Vaccine Sub-study: Percentage of Participants With Anti-tetanus Antibody Level >=0.1 IU/mL at Month 1-Tdap Vaccination
Description: Percentage of participants with anti-tetanus antibody level >=0.1 IU/mL at Month 1 were reported in this outcome measure. Two-sided 95% CI was based on Clopper-Pearson exact method.
Time Frame: Month 1
Population: as for outcome 27
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Vaccine Sub-study: Tdap Vaccination
Number analyzed (Participants) | 16
Percentage of participants | 100 [79.4 to 100.0]

29. Secondary Outcome: Vaccine Sub-study: Percentage of Participants With >=4 Times Increase in Anti-tetanus Antibody Level From Baseline at Month 1-Tdap Vaccination
Description: Percentage of participants with >=4 times increase in anti-tetanus antibody level from baseline were reported in this outcome measure. Two-sided 95% CI was based on Clopper-Pearson exact method.
Time Frame: Month 1
Population: as for outcome 27
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Vaccine Sub-study: Tdap Vaccination
Number analyzed (Participants) | 16
Percentage of participants | 50 [24.7 to 75.3]

30. Secondary Outcome: Vaccine Sub-study: Geometric Mean Fold Change in Anti-tetanus Levels Above Baseline Values at Month 1-Tdap Vaccination
Description: Geometric mean and 95% CI were calculated by exponentiating the mean logarithm of the observed data and the corresponding CIs. Fold change was defined as the ratio of the post-baseline result to the baseline result. The assay results below the LLOQ were set to 0.5 * LLOQ except when pre-vaccination assay results is < LLOQ while postvaccination result is >= LLOQ, in which case the pre-vaccination value will be set to LLOQ.
Time Frame: From Baseline (pre-vaccination on Day 1) to Month 1
Population: as for outcome 27
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | Vaccine Sub-study: Tdap Vaccination
Number analyzed (Participants) | 16
Fold change | 5.7 [3.1 to 10.6]

31. Secondary Outcome: Vaccine Sub-study: Geometric Mean Concentrations (GMCs) of Anti-tetanus Antibody Levels at Month 1-Tdap Vaccination
Description: Geometric mean and 95% CI were calculated by exponentiating the mean logarithm of the observed data and the corresponding CIs. Assay results below the LLOQ were set to 0.5* LLOQ.
Time Frame: Month 1
Population: as for outcome 27
Measure: Geometric Mean (95% Confidence Interval); unit: milli-international units (mIU)/mL
Arm/Group | Vaccine Sub-study: Tdap Vaccination
Number analyzed (Participants) | 16
milli-international units (mIU)/mL | 8.4 [5.8 to 12.1]

32. Secondary Outcome: Vaccine Sub-study: Percentage of Participants With Human Serum Bactericidal Activity (hSBA) Titer >=1:8 at Month 1 Post-vaccination for Serogroup C-Meningococcal ACWY Vaccination
Description: Percentage of participants with hSBA titer >=1.8 at 1 month post vaccination for serogroup C were reported in this outcome measure. Two-sided 95% CI was based on Clopper-Pearson exact method.
Time Frame: Month 1
Population: FAS-ACWY was defined as all participants who received the meningococcal ACWY vaccine (with or without the Tdap vaccine). Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Vaccine Sub-study: Meningococcal ACWY Vaccination: Participants who have received atleast 6 months of treatment with PF-06651600 50mg QD in the study B7981032 were continued to receive the study intervention while participating in this vaccine sub-study. Eligible participants who received the meningococcal ACWY vaccine with or without the Tdap vaccine were enrolled in this sub-study.
Arm/Group | Vaccine Sub-study: Meningococcal ACWY Vaccination
Number analyzed (Participants) | 5
Percentage of Participants | 20 [0.5 to 71.6]

33. Secondary Outcome: Vaccine Sub-study: Percentage of Participants With hSBA Titer >=1:4 at Month 1 Post-vaccination for Serogroup C-Meningococcal ACWY Vaccination
Description: Percentage of participants with hSBA titer >=1.4 at 1 month post vaccination for serogroup C were reported in this outcome measure. Two-sided 95% CI was based on Clopper-Pearson exact method.
Time Frame: Month 1
Population: as for outcome 32
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Vaccine Sub-study: Meningococcal ACWY Vaccination
Number analyzed (Participants) | 5
Percentage of Participants | 40 [5.3 to 85.3]

34. Secondary Outcome: Vaccine Sub-study: Geometric Mean Titers (GMT) of Antibodies for Serogroup C at Baseline and Month 1-Meningococcal ACWY Vaccination
Description: as for outcome 31
Time Frame: Baseline (pre-vaccination on Day 1) and Month 1
Population: as for outcome 32
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Vaccine Sub-study: Meningococcal ACWY Vaccination
Number analyzed (Participants) | 12
Titers
  Baseline | 5.7 [3.6 to 8.8]
  Month 1: number analyzed (Participants) | 11
  Month 1 | 14.1 [4.4 to 44.8]

35. Secondary Outcome: Vaccine Sub-study: Number of Participants With SAEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An SAE was any untoward medical occurrence that at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life-threatening; resulted in persistent disability/incapacity; was a congenital anomaly/birth defect; other important medical events.
Time Frame: From day of vaccination (Day 1) up to 35 days post last dose of vaccine (up to Day 36)
Population: SAS was defined as all participants from the vaccine sub study who received at least 1 vaccine (Tdap or meningococcal ACWY).
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine Sub-study: Tdap Vaccination | Vaccine Sub-study: Meningococcal ACWY Vaccination
Number analyzed (Participants) | 17 | 13
Participants | 0 | 0

36. Secondary Outcome: Vaccine Sub-study: Number of Participants With AEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: From day of vaccination (Day 1) up to 35 days post last dose of vaccine (up to Day 36)
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine Sub-study: Tdap Vaccination | Vaccine Sub-study: Meningococcal ACWY Vaccination
Number analyzed (Participants) | 17 | 13
Participants | 3 | 1

37. Secondary Outcome: Vaccine Sub-study: Number of Participants With AEs Leading to Discontinuation
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. AEs leading to discontinuation included participants who had an AE record that indicated that the AE caused the participant to be discontinued from the study or that action taken with study treatment was drug withdrawn.
Time Frame: From day of vaccination (Day 1) up to 35 days post last dose of vaccine (up to Day 36)
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine Sub-study: Tdap Vaccination | Vaccine Sub-study: Meningococcal ACWY Vaccination
Number analyzed (Participants) | 17 | 13
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Main Study: From start of study intervention (Day 1) until follow-up visit (4 weeks after last dose in Treatment period 1) (Up to Month 40). Vaccine Sub-study: From day of vaccination (Day 1) up to 35 days post last dose of vaccine (up to Day 36)
Description: For all-cause mortality, FAS was used. SAS was defined as all participants who took at least 1 dose of study intervention in the main study or sub-study. Same event may appear as both non-SAE and SAE but are distinct events. An event may be categorized as serious in 1 participant and non-serious in another, or a participant may have experienced both SAE and non-SAE.
Arm/Group | Main Study: Ritlecitinib 200 mg/ 50 mg QD (de Novo Participants) | Main Study: Ritlecitinib 50 mg QD (Roll-over Participants) | Vaccine Sub-study: Tdap Vaccination | Vaccine Sub-study: Meningococcal ACWY Vaccination
All-Cause Mortality (participants affected / at risk) | 1/447 | 1/603 | 0/17 | 0/13
Serious Adverse Events (participants affected / at risk) | 33/447 | 43/603 | 0/17 | 0/13
Other Adverse Events (participants affected / at risk) | 309/447 | 372/603 | 3/17 | 1/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Main Study: Ritlecitinib 200 mg/ 50 mg QD (de Novo Participants) (N=447) | Main Study: Ritlecitinib 50 mg QD (Roll-over Participants) (N=603) | Vaccine Sub-study: Tdap Vaccination (N=17) | Vaccine Sub-study: Meningococcal ACWY Vaccination (N=13)
Acute myocardial infarction (Cardiac disorders) | 3 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Blindness (Eye disorders) | 0 | 1 | 0 | 0
Retinal artery occlusion (Eye disorders) | 1 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0
Cyst rupture (General disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 2 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 2 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 4 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 1 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 1 | 0 | 0
Latent tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0 | 0
Pelvic abscess (Infections and infestations) | 1 | 0 | 0 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Vulval abscess (Infections and infestations) | 1 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Borderline mucinous tumour of ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Solitary fibrous tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bell's palsy (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 2 | 0 | 0
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Bipolar I disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Cervical polyp (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Miscarriage of partner (Social circumstances) | 1 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0 | 0
Varicose vein (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Main Study: Ritlecitinib 200 mg/ 50 mg QD (de Novo Participants) (N=447) | Main Study: Ritlecitinib 50 mg QD (Roll-over Participants) (N=603) | Vaccine Sub-study: Tdap Vaccination (N=17) | Vaccine Sub-study: Meningococcal ACWY Vaccination (N=13)
Diarrhoea (Gastrointestinal disorders) | 24 | 25 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 27 | 27 | 0 | 0
Fatigue (General disorders) | 47 | 41 | 0 | 0
Pyrexia (General disorders) | 59 | 64 | 0 | 0
COVID-19 (Infections and infestations) | 55 | 99 | 0 | 0
Folliculitis (Infections and infestations) | 21 | 32 | 0 | 0
Nasopharyngitis (Infections and infestations) | 62 | 65 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 56 | 73 | 0 | 0
Urinary tract infection (Infections and infestations) | 35 | 36 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
SARS-CoV-2 test positive (Investigations) | 108 | 127 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 21 | 33 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 98 | 93 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 46 | 74 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 28 | 16 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 44 | 59 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 57 | 38 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 41 | 29 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (3):
  • Study Protocol (2022-03-28): https://cdn.clinicaltrials.gov/large-docs/57/NCT04006457/Prot_003.pdf
  • Statistical Analysis Plan: Main study (2024-04-12): https://cdn.clinicaltrials.gov/large-docs/57/NCT04006457/SAP_004.pdf
  • Statistical Analysis Plan: sub study SAP (2023-06-20): https://cdn.clinicaltrials.gov/large-docs/57/NCT04006457/SAP_005.pdf